CLINICAL TRIAL: NCT03843645
Title: The Effect of General Versus Regional Anesthesia on Postoperative Sleep Quality
Brief Title: General Versus Regional Anesthesia and Postoperative Sleep Quality
Acronym: AnesthSleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Associate Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AnesthSleep
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Surgery; Sleep Disturbance; Sleep Disorder; Sleep Fragmentation; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Sleep
Keywords: anesthesia, general; anesthesia, regional; sleep disorder; REM stage
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders; Sleep Deprivation; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders | interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator completing the questionnaires will not be aware of patient group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia group (Active Comparator): patients allocated to the general anesthesia group will be subjected to general anesthesia with sevoflurane (inhalational agent) used for maintenance
  Interventions: Procedure: general anesthesia
- regional anesthesia group (Active Comparator): patients allocated to the regional anesthesia group will be subjected to combined spinal-epidural anesthesia with ropivacaine and fentanyl
  Interventions: Procedure: regional anesthesia

INTERVENTIONS:
Procedure: general anesthesia — surgical procedure under general anesthesia
  Arms: general anesthesia group
Procedure: regional anesthesia — surgical procedure under regional anesthesia
  Arms: regional anesthesia group

SUMMARY:
Major surgery can lead to postoperative disturbances in sleep patterns with subjective deterioration of sleep quality according to patients' reports as well as objective alterations of sleep architecture, as recorded by polysomnography Factors implicated in postoperative sleep disturbances include but are not limited to the severity of the surgical procedure, the neuroendocrine response to surgery, inadequate treatment of postoperative pain and external factors interfering with sleep, such as light, noise and therapeutic procedures There are no adequate data from current literature as to whether regional anesthesia is superior to general anesthesia regarding postoperative sleep quality in patients subjected to either mode of anesthesia. So, the aim of this study will be to assess the effect of two different anesthetic techniques (general versus regional) in patients subjected to similar operations Patients will be assessed with the Pittsburgh Sleep Quality Questionnaire (PSQI), regarding preoperative and long term postoperative sleep quality and sleep diaries regarding early postoperative sleep quality

DETAILED DESCRIPTION:
Major surgery can lead to postoperative disturbances in sleep patterns with subjective deterioration of sleep quality according to patients' reports as well as objective alterations of sleep architecture, as recorded by polysomnography.

These disturbances include severe sleep fragmentation, rapid eye movement (REM) and slow wave sleep significant reductions in duration as well as an increase in non-REM sleep stages. Spontaneous awakenings are also frequently reported.

After the third or fourth postoperative day, there is a substantial rebound in total REM activity, with frequent reports of vivid nightmares.

Factors implicated in postoperative sleep disturbances include but are not limited to the severity of the surgical procedure, the neuroendocrine response to surgery, inadequate treatment of postoperative pain and external factors interfering with sleep, such as light, noise and therapeutic procedures.

There are no adequate data from current literature as to whether regional anesthesia is superior to general anesthesia regarding postoperative sleep quality in patients subjected to either mode of anesthesia. There have been a few studies evaluating the effect of regional anesthesia on postoperative sleep quality after orthopedic procedures, without however comparing regional to general anesthesia in this setting. preliminary data from these studies suggest that regional anesthesia can also lead to postoperative sleep disturbances during the first postoperative nights, such as causing a reduction of REM stage.

So, the aim of this study will be to assess the effect of two different anesthetic techniques (general versus regional) in patients subjected to a similar operative procedure (saphenectomy).

Patients taking part in the study will be evaluated regarding their preoperative sleep quality by the Pittsburgh Sleep Quality Questionnaire (PSQI). The PSQI examines seven components of sleep quality retrospectively over a period of four weeks: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. The patient self-rates each of these seven areas of sleep. Scoring of answers is based on a 0-3 scale, whereby '3' reflects the negative extreme on the Likert scale. The global score is generated by summing up all seven component scores and ranges from 0 to 21, with higher values corresponding to reduced sleep quality.

Consequently, patients will be randomized to one of two groups: one group subjected to general anesthesia (maintenance with sevoflurane) and a second group subjected to combined spinal-epidural anesthesia Patients will be assessed postoperatively with sleep diaries regarding potential sleep disturbances while they will be subjected to a long-term assessment of sleep quality by the use of the PSQI one and three months postoperatively.

The clinical implications of this study lie in the fact that postoperative sleep disturbances can lead to postoperative hemodynamic instability, episodic hypoxemia and mental status deterioration, which can all untowardly affect the short and long-term postoperative outcome. It would be interesting to determine whether one of the two anesthetic regimes is superior to the other as far as postoperative disturbances in sleep architecture are concerned

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, American Society of Anesthesiologists (ASA) distribution I-III, scheduled for saphenectomy

Exclusion Criteria:

* Alcoholism
* Mental disability
* Psychiatric disease (depression, dementia)
* Preoperative use of sleeping medication
* Language barriers
* Lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
subjective sleep quality (evaluated by Pittsburgh Sleep Quality Index) | preoperative status, one month postoperatively
  change from preoperative status of subjective sleep quality (evaluated by Pittsburgh Sleep Quality Index) at one month postoperatively
subjective sleep quality (evaluated by Pittsburgh Sleep Quality Index) | preoperative status, three months postoperatively
  change from preoperative status of subjective sleep quality (evaluated by Pittsburgh Sleep Quality Index) at three months postoperatively

SECONDARY OUTCOMES:
sleep diary | first postoperative week
  subjective evaluation of sleep quality by patients, based on a sleep questionnaire (evaluation of sleep duration, number of nocturnal awakenings and marking of sleep quality)

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, Principal Investigator — Aretaieion University Hospital, Faculty of Medicine, University of Athens
Locations (1):
- Aretaieion University Hospital, Athens, Greece

REFERENCES:
- [Background] Rosenberg-Adamsen S, Kehlet H, Dodds C, Rosenberg J. Postoperative sleep disturbances: mechanisms and clinical implications. Br J Anaesth. 1996 Apr;76(4):552-9. doi: 10.1093/bja/76.4.552. No abstract available. PMID 8652329
- [Background] Aurell J, Elmqvist D. Sleep in the surgical intensive care unit: continuous polygraphic recording of sleep in nine patients receiving postoperative care. Br Med J (Clin Res Ed). 1985 Apr 6;290(6474):1029-32. doi: 10.1136/bmj.290.6474.1029. PMID 3921096
- [Background] Lehmkuhl P, Prass D, Pichlmayr I. General anesthesia and postnarcotic sleep disorders. Neuropsychobiology. 1987;18(1):37-42. doi: 10.1159/000118390. PMID 3444524
- [Background] Knill RL, Moote CA, Skinner MI, Rose EA. Anesthesia with abdominal surgery leads to intense REM sleep during the first postoperative week. Anesthesiology. 1990 Jul;73(1):52-61. doi: 10.1097/00000542-199007000-00009. PMID 2360740
- [Background] Brimacombe J, Macfie AG. Peri-operative nightmares in surgical patients. Anaesthesia. 1993 Jun;48(6):527-9. doi: 10.1111/j.1365-2044.1993.tb07078.x. PMID 8322996
- [Background] Libert JP, Bach V, Johnson LC, Ehrhart J, Wittersheim G, Keller D. Relative and combined effects of heat and noise exposure on sleep in humans. Sleep. 1991 Feb;14(1):24-31. doi: 10.1093/sleep/14.1.24. PMID 1811316
- [Background] Dette F, Cassel W, Urban F, Zoremba M, Koehler U, Wulf H, Graf J, Steinfeldt T. Occurrence of rapid eye movement sleep deprivation after surgery under regional anesthesia. Anesth Analg. 2013 Apr;116(4):939-43. doi: 10.1213/ANE.0b013e3182860e58. Epub 2013 Mar 4. PMID 23460574
- [Background] Krenk L, Jennum P, Kehlet H. Sleep disturbances after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Nov;109(5):769-75. doi: 10.1093/bja/aes252. Epub 2012 Jul 24. PMID 22831887
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Reeder MK, Muir AD, Foex P, Goldman MD, Loh L, Smart D. Postoperative myocardial ischaemia: temporal association with nocturnal hypoxaemia. Br J Anaesth. 1991 Nov;67(5):626-31. doi: 10.1093/bja/67.5.626. PMID 1751279
- [Background] Rosenberg J, Wildschiodtz G, Pedersen MH, von Jessen F, Kehlet H. Late postoperative nocturnal episodic hypoxaemia and associated sleep pattern. Br J Anaesth. 1994 Feb;72(2):145-50. doi: 10.1093/bja/72.2.145. PMID 8110563
- [Background] Horne JA. Sleep loss and "divergent" thinking ability. Sleep. 1988 Dec;11(6):528-36. doi: 10.1093/sleep/11.6.528. PMID 3238256